CLINICAL TRIAL: NCT02866331
Title: Phase II, Randomized, Double-blind Clinical Trial for Efficacy of G-CSF and Autologous Cord Blood Infusion in Children With Cerebral Palsy
Brief Title: G-CSF and Autologous Cord Blood Infusion in Cerebral Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanyang University Seoul Hospital (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Young-Ho Lee, Professor, Department of Pediatrics, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-CB-G-2016
Record Dates: First submitted 2016-07-26; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Granulocyte Colony-Stimulating Factor; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CB + G-CSF (Experimental)
  Interventions: Drug: G-CSF (Leucostim); Biological: CB (autologous cord blood)
- CB + placebo (Placebo Comparator)
  Interventions: Biological: CB (autologous cord blood); Drug: Placebo (Normal saline)
- G-CSF (Experimental)
  Interventions: Drug: G-CSF (Leucostim)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Normal saline)

INTERVENTIONS:
Drug: G-CSF (Leucostim)
  Arms: CB + G-CSF; G-CSF
Biological: CB (autologous cord blood)
  Arms: CB + G-CSF; CB + placebo
Drug: Placebo (Normal saline)
  Arms: CB + placebo; Placebo

SUMMARY:
This study is performed to reveal the safety and feasibility of combination therapy with autologous cord blood mononuclear cells (CB) and G-CSF as well as repeated administration of G-CSF for children with cerebral palsy. The evaluation tools are as follows: (1) Developmental tests (DDST, PEDI, GMFM, GMFCS, MACS, QUEST), (2) Neurocognitive function test (WPPSI-IV), (3) Brain MRI-DTI, (4) Peripheral blood CD34+ cell counts, (5) Neurotrophic factors/anti-inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Ages from 2 years to 10 years at the time of enrollment
* Non-severe type of cerebral palsy
* Willing to comply with all study procedures

Exclusion Criteria:

* Previous participation within 1 year in a clinical study with stem cell therapy including cord blood, G-CSF, and erythropoietin
* Presence of chromosomal abnormalities
* Unwillingness to participate clinical trial
* Presence of hypersensitivity reaction to G-CSF
* Evidence of hepatic, renal, cardiac dysfunctions

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Confirm the safety of autologous cord blood infusion and repeated injection of G-CSF in children with cerebral palsy by repeated follow-up every 3 months over 18 months with clinical and laboratory evaluations | For 18 months from date of randomization

SECONDARY OUTCOMES:
Confirm the efficacy of autologous cord blood infusion and/or G-CSF in children with cerebral palsy using standardized Gross Motor Function Measure evaluation. | Every 6 months from date of randomization up to 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes